CLINICAL TRIAL: NCT04853745
Title: Analyzing the Effect of Different Polishing Materials on Different Dental Tissues by Micro-Computed Tomography
Brief Title: The Effect of Air Polishing on the Tooth Surface
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Vecihe Merve Balta Uysal, research assistant, Kocaeli University
Other Study IDs: KOU GOKAEK 2019/10.34
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dental Plaque
Keywords: glycine; erythritol; sodium bicarbonate; x-ray microtomography; gingival recession; air abrasion
MeSH Terms: conditions — Dental Plaque; Gingival Recession

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- sodium bicarbonate group: Sodium bicarbonate-based powder (CLASSIC®, EMS SA, Nyon, Switzerland) was used for air polishing the samples belonging to this group. All surfaces were numbered and application was made to the mesial and distal surfaces of the root, buccal and lingual surfaces of the crown to avoid repeated instrumentations. After device and samples were fixed, a metal plate with a 5 mm diameter hole was placed on the sample to limit the application area. Surfaces one and three were air-polished using the with a medium power setting (9 LED power setting), and surfaces two and four were air-polished using the with a maximum power setting (17 LED power setting). The distance between the handpiece and the tooth surface was kept constant at 5 mm, and the treatment angulation was adjusted to 60 degrees. In all applications, the application time was 5 seconds and the water setting was medium (6 LED). The powder chambers of the device were filled to the maximum level in each application.
  Interventions: Device: AIR-FLOW® Master Piezon
- glycine group: Glycine-based powder (PERIO®, EMS SA, Nyon, Switzerland) was used for air polishing the samples belonging to this group. All surfaces were numbered and application was made to the mesial and distal surfaces of the root, buccal and lingual surfaces of the crown to avoid repeated instrumentations. After device and samples were fixed, a metal plate with a 5 mm diameter hole was placed on the sample to limit the application area. Surfaces one and three were air-polished using the with a medium power setting (9 LED power setting), and surfaces two and four were air-polished using the with a maximum power setting (17 LED power setting). The distance between the handpiece and the tooth surface was kept constant at 5 mm, and the treatment angulation was adjusted to 60 degrees. In all applications, the application time was 5 seconds and the water setting was medium (6 LED). The powder chambers of the device were filled to the maximum level in each application.
  Interventions: Device: AIR-FLOW® Master Piezon
- erythritol group: Erythritol-based powder (PLUS®, EMS SA, Nyon, Switzerland) was used for air polishing the samples belonging to this group. All surfaces were numbered and application was made to the mesial and distal surfaces of the root, buccal and lingual surfaces of the crown to avoid repeated instrumentations. After device and samples were fixed, a metal plate with a 5 mm diameter hole was placed on the sample to limit the application area. Surfaces one and three were air-polished using the with a medium power setting (9 LED power setting), and surfaces two and four were air-polished using the with a maximum power setting (17 LED power setting). The distance between the handpiece and the tooth surface was kept constant at 5 mm, and the treatment angulation was adjusted to 60 degrees. In all applications, the application time was 5 seconds and the water setting was medium (6 LED). The powder chambers of the device were filled to the maximum level in each application.
  Interventions: Device: AIR-FLOW® Master Piezon

INTERVENTIONS:
Device: AIR-FLOW® Master Piezon — AIR-FLOW® Master Piezon is intended for use in the cleaning and polishing of teeth by the projection of water,air, and dental powders onto the tooth surface. The device removes dental plaque, soft deposits, and surface stains from pits, grooves, interproximal spaces, or smooth surfaces of teeth. This air polishing device was used for all powder instrumentations.

SUMMARY:
The use of air-polishing device that operates by directing a fine slurry of pressurized air, water, and abrasive particles has become widespread in dentistry for polishing. The introduction of abrasive powders with different properties creates the need to evaluate the effects of these powders on dental hard tissues. This study was focused on the effect of sodium bicarbonate, glycine and erythritol air polishing on enamel and exposed root surface.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of sodium bicarbonate, glycine and erythritol air polishing on enamel and exposed root surface. Forty eight single root extracted teeth were included into the study. The teeth were divided into three groups, the crown and exposed root surface were air polished using three powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) at baseline and then after powder treatment and the defect depth, defect volume, demineralization depth and mineral density values were estimated.

ELIGIBILITY:
Inclusion Criteria:

* Being older than age of 18,
* Willing to participate the study,
* To have a single rooted tooth with gingival recession on all surfaces and need to be extracted,
* The tooth has to be free of caries, defects and restorations.

Exclusion Criteria:

Have history of infectious diseases like Hepatitis and/or HIV (+).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were recruited from individuals seeking periodontal and/or dental treatment at Kocaeli University, Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Defect depth | 5 second
  The teeth were divided into three groups, the crown and exposed root surface were air polished using three powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) at baseline and then after powder treatment and the defect depth was estimated.
Demineralization depth | 5 second
  The teeth were divided into three groups, the crown and exposed root surface were air polished using three powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) at baseline and then after powder treatment and the demineralization depth was estimated.
Mineral density | 10 second
  The teeth were divided into three groups, the crown and exposed root surface were air polished using three powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5 mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) at baseline and then after powder treatment and the mineral density was estimated.
Defect volume | 5 second
  The teeth were divided into three groups, the crown and exposed root surface were air polished using three powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) at baseline and then after powder treatment and the defect volume was estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Faculty of Dentistry, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petersilka GJ. Subgingival air-polishing in the treatment of periodontal biofilm infections. Periodontol 2000. 2011 Feb;55(1):124-42. doi: 10.1111/j.1600-0757.2010.00342.x. No abstract available. PMID 21134232
- [Background] Graumann SJ, Sensat ML, Stoltenberg JL. Air polishing: a review of current literature. J Dent Hyg. 2013 Aug;87(4):173-80. PMID 23986410
- [Background] Gutmann ME. Air polishing: a comprehensive review of the literature. J Dent Hyg. 1998 Summer;72(3):47-56. PMID 9693568
- [Background] Weaks LM, Lescher NB, Barnes CM, Holroyd SV. Clinical evaluation of the Prophy-Jet as an instrument for routine removal of tooth stain and plaque. J Periodontol. 1984 Aug;55(8):486-8. doi: 10.1902/jop.1984.55.8.486. PMID 6592321
- [Background] Berkstein S, Reiff RL, McKinney JF, Killoy WJ. Supragingival root surface removal during maintenance procedures utilizing an air-powder abrasive system or hand scaling. An in vitro study. J Periodontol. 1987 May;58(5):327-30. doi: 10.1902/jop.1987.58.5.327. PMID 3295185
- [Background] Barnes CM, Russell CM, Gerbo LR, Wells BR, Barnes DW. Effects of an air-powder polishing system on orthodontically bracketed and banded teeth. Am J Orthod Dentofacial Orthop. 1990 Jan;97(1):74-81. doi: 10.1016/S0889-5406(05)81712-3. No abstract available. PMID 2136972
- [Background] Kontturi-Narhi V, Markkanen S, Markkanen H. Effects of airpolishing on dental plaque removal and hard tissues as evaluated by scanning electron microscopy. J Periodontol. 1990 Jun;61(6):334-8. doi: 10.1902/jop.1990.61.6.334. PMID 2366141
- [Background] Atkinson DR, Cobb CM, Killoy WJ. The effect of an air-powder abrasive system on in vitro root surfaces. J Periodontol. 1984 Jan;55(1):13-8. doi: 10.1902/jop.1984.55.1.13. PMID 6319658
- [Background] Barnes CM, Covey D, Watanabe H, Simetich B, Schulte JR, Chen H. An in vitro comparison of the effects of various air polishing powders on enamel and selected esthetic restorative materials. J Clin Dent. 2014;25(4):76-87. PMID 26054183
- [Background] Pelka M, Trautmann S, Petschelt A, Lohbauer U. Influence of air-polishing devices and abrasives on root dentin-an in vitro confocal laser scanning microscope study. Quintessence Int. 2010 Jul-Aug;41(7):e141-8. PMID 20614037
- [Background] Sahrmann P, Ronay V, Schmidlin PR, Attin T, Paque F. Three-dimensional defect evaluation of air polishing on extracted human roots. J Periodontol. 2014 Aug;85(8):1107-14. doi: 10.1902/jop.2014.130629. Epub 2014 Jan 30. PMID 24476548
- [Background] Tada K, Kakuta K, Ogura H, Sato S. Effect of particle diameter on air polishing of dentin surfaces. Odontology. 2010 Feb;98(1):31-6. doi: 10.1007/s10266-009-0113-8. Epub 2010 Feb 16. PMID 20155505
- [Background] Tada K, Wiroj S, Inatomi M, Sato S. The characterization of dentin defects produced by air polishing. Odontology. 2012 Jan;100(1):41-6. doi: 10.1007/s10266-011-0019-0. Epub 2011 May 10. PMID 21556726
- [Background] Herr ML, DeLong R, Li Y, Lunos SA, Stoltenberg JL. Use of a continual sweep motion to compare air polishing devices, powders and exposure time on unexposed root cementum. Odontology. 2017 Jul;105(3):311-319. doi: 10.1007/s10266-016-0282-1. Epub 2017 Jan 9. PMID 28070701
- [Background] Camboni S, Donnet M. Tooth Surface Comparison after Air Polishing and Rubber Cup: A Scanning Electron Microscopy Study. J Clin Dent. 2016 Mar;27(1):13-18. PMID 28390211
- [Background] Petersilka GJ, Bell M, Mehl A, Hickel R, Flemmig TF. Root defects following air polishing. J Clin Periodontol. 2003 Feb;30(2):165-70. doi: 10.1034/j.1600-051x.2003.300204.x. PMID 12622860
- [Background] Petersilka GJ, Bell M, Haberlein I, Mehl A, Hickel R, Flemmig TF. In vitro evaluation of novel low abrasive air polishing powders. J Clin Periodontol. 2003 Jan;30(1):9-13. doi: 10.1034/j.1600-051x.2003.300102.x. PMID 12702105
- [Background] Agger MS, Horsted-Bindslev P, Hovgaard O. Abrasiveness of an air-powder polishing system on root surfaces in vitro. Quintessence Int. 2001 May;32(5):407-11. PMID 11444076
- [Background] Galloway SE, Pashley DH. Rate of removal of root structure by the use of the Prophy-Jet device. J Periodontol. 1987 Jul;58(7):464-9. doi: 10.1902/jop.1987.58.7.464. PMID 3476717